CLINICAL TRIAL: NCT04463901
Title: Intraoperative Mitomycin C Combined With Conjunctival Autograft or Limbal Conjunctival Autograft for Recurrent Pterygium: a Randomized Clinical Trial
Brief Title: Conjunctival Autograft or Limbal Conjunctival Autograft for Recurrent Pterygium Using Mitomycin C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shiyou Zhou, MD,PhD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20150527
Record Dates: First submitted 2020-07-04; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Recurrent Pterygium
Keywords: recurrent pterygium; pterygium; limbal conjunctival autograft; conjunctival autograft; mitomycin c
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group CAG (Active Comparator): After pterygium excision, intraoperative mitomycin c (0.02%) for 5 minutes will be applied topically onto the exposed surgical area and then conjunctival autograft without limbal tissue will be used to cover the bare sclera.
  Interventions: Procedure: Pterygium excision; Procedure: Intraoperative mitomycin C; Procedure: Conjunctival autograft
- Group LCAG (Active Comparator): After pterygium excision, intraoperative mitomycin c (0.02%) for 5 minutes will be applied topically onto the exposed surgical area and then limbal conjunctival autograft will be used to cover the bare sclera.
  Interventions: Procedure: Pterygium excision; Procedure: Intraoperative mitomycin C; Procedure: Limbal conjunctival autograft

INTERVENTIONS:
Procedure: Pterygium excision — Partial conjunctiva and anterior tenon's membrane underneath will be removed after the excision of pterygium tissue.
Procedure: Intraoperative mitomycin C — Intraoperative mitomycin C (0.02%) will be applied for 5 minutes after pterygium excision.
  Other Names: MMC
Procedure: Conjunctival autograft — A conjunctival autograft will be applied to cover the conjunctival defect after pterygium excision.
  Other Names: CAG
  Arms: Group CAG
Procedure: Limbal conjunctival autograft — A limbal conjunctival autograft will be applied to cover the conjunctival defect after pterygium excision.
  Other Names: LCAG
  Arms: Group LCAG

SUMMARY:
The purpose of this randomized clinical trial is to compare the efficacy and safety of intraoperative mitomycin C(MMC) combined with limbal conjunctival autograft(LCAG) or conjunctival autograft(CAG) for recurrent pterygium surgery. The investigators will also evaluate particular risk factors related to pterygium recurrence

DETAILED DESCRIPTION:
Intraoperative mitomycin C after pterygium excision is widely used to prevent recurrce of recurrent pterygium. Conjunctival autograft with or without limbal tissue used to cover the bare sclera will efficiently reduce postoperative longstanding epithelial defect.

Patients with recurrent pterygium will be randomly assigned to undertake pterygium excision followed by intraoperative mitomycin C with conjunctival autograft or limbal conjunctival autograft .The patients will be followed at least 12 months. Corneal recurrence is considered as a fibrovascular ingrowth beyond the limbus with conjunctival drag in the area of previous pterygium excision.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent pterygium
* Willingness to participate in research project and to attend research time
* At least 6 months after last pterygium surgery

Exclusion Criteria:

* Pregnant,breast-feeding women or poor general health
* Patients with significant ocular or lid pathology, such as Sjogren's Syndrome ,infection, exposure keratitis,glaucoma and trauma
* Patients with allergy to mitomycin C,tobramycin or local anesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2016-02; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Recurrence of pterygium | One year

SECONDARY OUTCOMES:
Visual acuity | One year
Healing time of corneal epithelium | Four weeks
Healing time of conjunctival epithelium | Four weeks
Postoperative complications | One year

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Shiyou, M.D., Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China